CLINICAL TRIAL: NCT05294055
Title: A Prospective and Multicenter Clinical Study of Mecapegfilgrastim in Combination With Chemotherapy for Autologous Peripheral Blood Stem Cell Mobilization in Patients With Multiple Myeloma or Lymphoma
Brief Title: Mecapegfilgrastim With Chemotherapy for Peripheral Blood Stem Cell Mobilization in MM and Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Jiangsu Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2021036
Record Dates: First submitted 2022-03-15; First posted 2022-03-24 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Multiple Myeloma; Lymphoma
Keywords: peripheral blood stem cell mobilization; Mecapegfilgrastim; chemotherapy
MeSH Terms: conditions — Multiple Myeloma; Lymphoma | interventions — Etoposide; Cyclophosphamide; pegylated granulocyte colony-stimulating factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- lymphoma, chemotherapy plus Mecapegfilgrastim SC on day 2 (Experimental)
  Interventions: Drug: Etoposide; Drug: Mecapegfilgrastim, day 2
- lymphoma, chemotherapy plus Mecapegfilgrastim SC on day 5 (Experimental)
  Interventions: Drug: Etoposide; Drug: Mecapegfilgrastim, day 5
- myltiple myeloma, chemotherapy plus Mecapegfilgrastim SC on day 2 (Experimental)
  Interventions: Drug: Cyclophosphamide; Drug: Mecapegfilgrastim, day 2
- myltiple myeloma, chemotherapy plus Mecapegfilgrastim SC on day 5 (Experimental)
  Interventions: Drug: Cyclophosphamide; Drug: Mecapegfilgrastim, day 5

INTERVENTIONS:
Drug: Etoposide — Etoposide 1.5-1.8g/m2, single dose
  Arms: lymphoma, chemotherapy plus Mecapegfilgrastim SC on day 2; lymphoma, chemotherapy plus Mecapegfilgrastim SC on day 5
Drug: Cyclophosphamide — Cyclophosphamide 50mg/kg or 2g/m2, for 2 days
  Arms: myltiple myeloma, chemotherapy plus Mecapegfilgrastim SC on day 2; myltiple myeloma, chemotherapy plus Mecapegfilgrastim SC on day 5
Drug: Mecapegfilgrastim, day 2 — Mecapegfilgrastim 12mg SC, on day 2 after chemotherapy
  Arms: lymphoma, chemotherapy plus Mecapegfilgrastim SC on day 2; myltiple myeloma, chemotherapy plus Mecapegfilgrastim SC on day 2
Drug: Mecapegfilgrastim, day 5 — Mecapegfilgrastim 12mg SC, on day 5 after chemotherapy
  Arms: lymphoma, chemotherapy plus Mecapegfilgrastim SC on day 5; myltiple myeloma, chemotherapy plus Mecapegfilgrastim SC on day 5

SUMMARY:
This is a multicenter prospective study to evaluate the efficacy and safety of chemotherapy combined with a single dose of subcutaneous(SC) injection mecapegfilgrastim on day 2 or day 5 after chemotherapy for autologous peripheral blood stem cell (PBSC) mobilization in patients with multiple myeloma or lymphoma.

DETAILED DESCRIPTION:
Subjects eligible for autologous stem-cell transplantation are randomized to receive a single dose of 12mg mecapegfilgrastim SC on day 2 or day 5 after chemotherapy for PBSC mobilization. According to the protocol, high-dose cyclophosphamide (50mg/kg or 2g/m2, for 2 days) is given to patients with MM, and high-dose etoposide (1.5-1.8g/m2, single dose ) is administered to patients with lymphoma. Apheresis is performed according to the standard institutional regulations. The primary point is to evaluate the percentage of successful mobilization, defined as the cumulative collection of ≥2×10^6/kg CD34+ cells in three or fewer apheresis.

ELIGIBILITY:
Inclusion Criteria:

1. Lymphoma patients with ≤2 lines of prior therapy, patients with multiple myeloma with one line of therapy;
2. Patients who had achieved at least partial response (PR);
3. Patients who were eligible for autologous peripheral blood stem cell transplantation
4. Age≥18 and≤65 years;
5. Patients with Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
6. Patients who have an estimated life expectancy of more than three months
7. Fertile patients must be willing to use reliable contraception during the clinical study period and for 90 days after the last dose and have a negative serological pregnancy test within 72 hours prior to the first dose.
8. Patients must be able and willing to give written informed consent prior to any study-related procedures

Exclusion Criteria:

1. Patients who had previously attempted hematopoietic stem cell mobilization;
2. Patients who had undergone previous bone marrow transplantation;
3. Lymphoma patients with bone marrow involvement or patients with MM who had >10% bone marrow involvement at screening ;
4. Patients with angina pectoris, myocardial infarction, coronary stent implantation, uncontrolled arrhythmias (atrial tachycardia, atrial fibrillation, persistent ventricular arrhythmias, etc.), cardiac insufficiency, Q-Tc interval >500ms, left ventricular ejection fraction (EF)<60%, or other heart diseases that the investigator considers unsuitable for hematopoietic stem cell mobilization or hematopoietic stem cell transplantation;
5. Patients with uncontrolled pulmonary infection;
6. Patients who had any of the following laboratory indicators:

   1. White blood cell count(WBC)<2.5×109/L；
   2. Absolute neutrophil count(ANC)<1.5×109/L；
   3. Platelets count(PLT)<80×109/L；
   4. Creatinine > 2.0 X ULN of the reference range or creatinine clearance ≤60ml/min
   5. AST/ALT/Total bilirubin > 2.5 X ULN；
7. Patients who have received any of the following treatments:

   1. Patients who had been treated with more than 4 cycles of lenalidomide or received lenalidomide within 4 weeks prior to hematopoietic stem cell mobilization chemotherapy.
   2. Patients who previously been treated with fludarabine or melphalan;
   3. Patients who plan to receive radiation within 30 days after transplantation
   4. Patients who had received radiation therapy in the pelvis
8. Patients allergic to Mecapegfilgrastim, pegylated granulocyte stimulating factor, granulocyte stimulating factor, or other formulations expressed by E. coli.
9. Patients who are pregnant or breastfeeding
10. Patients who are participating in other clinical studies or the interval of the last dose of prior study drug to the mobilization chemotherapy is less than 4 weeks (or 5 half-lives of the study drug);
11. Patients with other conditions unsuitable for this study according to the investigator's judgment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-04-26 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
percentage of successful mobilization | up to 28 days since the last subject were given mecapegfilgrastim
  The percentage of subjects with ≥2×106 cell/kg CD34+ cells were collected.

SECONDARY OUTCOMES:
the number of the total CD34+ cells | up to 28 days since the last subject were given mecapegfilgrastim
  the number of the total CD34+ cells which were collected from each subject
the number of leukaphereses | up to 28 days since the last subject were given mecapegfilgrastim
  the number of leukaphereses needed to collect ≥2×10^6/kg CD34+ cells
Incidence of febrile neutropenia (FN) | up to 28 days since the last subject were given mecapegfilgrastim
  incidence of FN during chemotherapy plus mecapegfilgrastim mobilization
times to neutrophil and platelet engraftment | up to 1 year post-transplantation
  times to neutrophil and platelet engraftment after autologous stem cell transplantation

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Shandong Cancer Hospital, Jinan, Shandong
  - Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No